CLINICAL TRIAL: NCT03002389
Title: Hyperpolarized Xenon-129 MRI: a New Multi-dimensional Biomarker to Determine Pulmonary Physiologic Responses to COPD Therapeutics
Status: Active, not recruiting | Phase: Phase 2 | Type: Interventional
Sponsor: University of Virginia (Other)
Responsible Party: Principal Investigator, Y. Michael Shim, MD, Assoicate Professor, Department of Medicine, University of Virginia
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Diagnostic
Other Study IDs: 19569-19352
Record Dates: First submitted 2016-12-13; First posted 2016-12-23 (Estimated); Last update posted 2024-11-18 (Actual); Status verified 2024-11

CONDITIONS: Chronic Obstructive Pulmonary Disease
Keywords: chronic obstructive pulmonary disease; COPD; emphysema; MRI; hyper polarized gas MRI
MeSH Terms: conditions — Pulmonary Disease, Chronic Obstructive; Emphysema | interventions — GSK573719; vilanterol; Fluticasone

STUDY DESIGN:
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: Yes | FDA-regulated Device: No

ARMS (1):
- All COPD Subjects (Other): All subjects will be assessed with hyper polarized xenon-129 MRI, pulmonary function test, quality of life measures (BDI, TDI, SGRQ, CRQ, BODE, GOLD), and blood test.
  Intervention: All subjects will received Anoro one puff once a day for 30 days first, then 3 day washout, then Arnuity 250 microgram one puff twice a day for 30 days to complete the study.
  Interventions: Drug: Anoro Ellipta; Drug: Arnuity Ellipta

INTERVENTIONS:
Drug: Anoro Ellipta — inhaler approved by FDA (strength umeclidinium 65 microgram + vilanterol 25 microgram) One puff once a day for 30 days
  Other Names: umeclidinium + vilanterol
Drug: Arnuity Ellipta — inhaler approved by FDA (strength 250 microgram) One puff twice a day for 30 days
  Other Names: fluticasone

SUMMARY:
Hyper polarized xenon-129 MRI (HXe MRI) is a unique imaging test which can detect how air is flowing in and out of lungs and how oxygen can move from inhaled air into the blood. Chronic Obstructive Pulmonary Disease (COPD) is a disease in which patients develop narrowing of airways, thus, having difficulties breathing air in and out their lungs and also damaging the lung tissues which patients need to move oxygen from the air into blood.

In this study, two drugs which are already approved by FDA (Anoro and Arnuity) will be administered to patients who are already known to have COPD. While patients are being treated with these two drugs (one drug at a time over a month), lung health by using usual testing methods (CT scan of the lung, pulmonary function test, and blood test) will be assessed in addition to HXe MRI.

The goal of this study is to prove that the HXe MRI is an excellent imaging test to show the state of lung health among COPD patients and also to obtain new informations on how lung health changes with drugs that are already approved by US FDA. This work is anticipated to help develop HXe MRI as a new clinical test which can guide how to treat patients with COPD and if new therapies can improve lung health of patients with COPD.

ELIGIBILITY:
Inclusion Criteria:

* post bronchodilator PFT spirometry FEV1/FVC < 70% predicted
* History of diagnosis of COPD
* History of alpha 1 anti-trypsin deficiency

Exclusion Criteria:

* previous diagnosis of asthma, interstitial lung disease, pulmonary vascular disease, inability to complete MRI or any of the assessment testings.

Ages: 18 Years to 85 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 95 (Estimated)
Dates: Start 2017-11-05 (Actual); Primary Completion 2023-12-31 (Actual); Study Completion 2028-01-31 (Estimated)

PRIMARY OUTCOMES:
Changes in the hyper polarized MRI xenon-129 MRI (HXe MRI) assessment pre-post 30-day treatment of umeclidinium+vilanterol or Flovent | Time point with +/- 7 day window: first baseline=day 0, first follow-up=day 30, second baseline=day 37, second follow-up=day 67
  In vivo lung physiology measurement obtained by HXe MRI pre and post drug intervention.
  In vivo lung physiology is measured by % of the lung that does not ventilate (dead space ventilation), among of the dissolved xenon-129 gas location among airways, interstitial tissues, or circulating red blood cells. These measures will be reported as continuous variables for data analyses.

SECONDARY OUTCOMES:
High resolution CT of lung | First baseline only=day 0
  Quantification of emphysematous lung tissues and abnormally thickened airways in correlation with changed detectable by HXe MRI.
  % of lung tissues with emphysema will be quantified by measuring tissue density using Hounsfield Unit (HU). Based on COPDgene and other studies, we will use HU < -950 as emphysematous lung tissue. The lung CT scan will then be processed to yield % of lung tissue with emphysema. The airway thickness will be measured by standardized imaging algorithm developed by VIDA imaging.
Changes in pulmonary Function Test (PFT) from pre to post-umeclidinium+vilanterol or Flovent | Time point with +/- 7 day window: first baseline=day 0, first follow-up=day 30, second baseline=day 37, second follow-up=day 67
  Measurement of in vivo lung physiology using clinical standard testing in correlation with HXe MRI changes pre and post drug intervention.
  The gas exchange capacity will be assessed by diffusion capacity of carbon monoxide represented as percent DLCO. This is a standard clinical measure being used routinely in pulmonary clinics.
Changes in Baseline Dyspnea Index from pre to post-umeclidinium+vilanterol or flovent | Time point with +/- 7 day window: first baseline=day 0, first follow-up=day 30, second baseline=day 37, second follow-up=day 67
  Measurement of in vivo lung physiology using clinical standard quality of life testing in correlation with HXe MRI changes pre and post drug intervention.
  Quality of life survey will be administered to obtain numeric number as a results.
Changes in Transient Dyspnea Index from pre to post-umeclidinium+vilanterol or flovent | Time point with +/- 3 day window: first baseline=day 0, first follow-up=day 30, second baseline=day 37, second follow-up=day 67
  Measurement of in vivo lung physiology using clinical standard quality of life testing in correlation with HXe MRI changes pre and post drug intervention.
  Quality of life survey will be administered to obtain numeric number as a results.
Changes in Saint George's Respiratory Questionnaire from pre to post-umeclidinium+vilanterol or flovent | Time point with +/- 3 day window: first baseline=day 0, first follow-up=day 30, second baseline=day 37, second follow-up=day 67
  Measurement of in vivo lung physiology using clinical standard quality of life testing in correlation with HXe MRI changes pre and post drug intervention.
  Quality of life survey will be administered to obtain numeric number as a results.
Changes in Chronic Respiratory Questionnaire from pre to post-umeclidinium+vilanterol or flovent | Time point with +/- 3 day window: first baseline=day 0, first follow-up=day 30, second baseline=day 37, second follow-up=day 67
  Measurement of in vivo lung physiology using clinical standard quality of life testing in correlation with HXe MRI changes pre and post drug intervention.
  Quality of life survey will be administered to obtain numeric number as a results.
Changes in BODE score from pre to post-umeclidinium+vilanterol or flovent | Time point with +/- 3 day window: first baseline=day 0, first follow-up=day 30, second baseline=day 37, second follow-up=day 67
  Measurement of in vivo lung physiology and mortality prediction score using clinical standard testing in correlation with HXe MRI changes pre and post drug intervention. BODE score is calculated by the results from the pulmonary function test, modified medical research council score, and body mass index. This will yield a score ranging from 0 to 10 with higher scores predicting higher chance of mortality.
Changes in GOLD Stage from pre to post-umeclidinium+vilanterol or flovent | Time point with +/- 3 day window: first baseline=day 0, first follow-up=day 30, second baseline=day 37, second follow-up=day 67
  Measurement of in vivo lung physiology and mortality prediction score using clinical standard testing in correlation with HXe MRI changes pre and post drug intervention.
  GOLD stage is calculated by a combination of pulmonary function test result, modified medical research council score, and history of frequency of COPD exacerbation previous 12 months. This score will yield GOLD stages A (mild) to , B, C, D (most severe).

CONTACTS AND LOCATIONS:
Overall Officials: Yun M Shim, MD, Principal Investigator — University of Virginia; Kun Qing, PhD, Principal Investigator — University of Virginia
Locations (1):
- Roselove NUNOO-ASARE, Keswick, Virginia, United States

IPD SHARING:
Plan to Share IPD: Undecided
At the conclusion of the study, correlation data between COPD phenotypes and changes in MRI characteristics will be shared. Data from individuals will be complied with unique study-generated subject ID after removing all personal identifiers. Once this is completed, the data may be shared with hyper polarized MR imaging network currently being formed in collaboration with University of WI, U Penn, Duke, U of Cincinnati, and U Missouri. The data will be accessible by these investigators after the data sharing plans are reviewed by the IRB of the record (at the University of Virginia).

REFERENCES:
- [Result] Qing K, Ruppert K, Jiang Y, Mata JF, Miller GW, Shim YM, Wang C, Ruset IC, Hersman FW, Altes TA, Mugler JP 3rd. Regional mapping of gas uptake by blood and tissue in the human lung using hyperpolarized xenon-129 MRI. J Magn Reson Imaging. 2014 Feb;39(2):346-59. doi: 10.1002/jmri.24181. Epub 2013 May 16. PMID 23681559
- [Result] Qing K, Mugler JP 3rd, Altes TA, Jiang Y, Mata JF, Miller GW, Ruset IC, Hersman FW, Ruppert K. Assessment of lung function in asthma and COPD using hyperpolarized 129Xe chemical shift saturation recovery spectroscopy and dissolved-phase MRI. NMR Biomed. 2014 Dec;27(12):1490-501. doi: 10.1002/nbm.3179. Epub 2014 Aug 22. PMID 25146558